CLINICAL TRIAL: NCT03723525
Title: Evaluation of World Health Organization (WHO) Recommendations on Test and Treat Strategy, Managing Advanced HIV Disease and Rapid Initiation of ART Among People Living With HIV in Nepal: A Cluster Randomized Trial.
Brief Title: Package of Care to Improve Retention in ART and Mortality Among Treatment Naive HIV Infected Individuals
Acronym: PRAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Centre for AIDs and STD Control, Nepal (Other Government)
Collaborators: Sukraraj Tropical and Infectious Disease Hospital (Unknown); National Academy of Medical Sciences, Nepal (Other Government); Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other); Rapti Sub-regional Hospital (Unknown); Western Regional Hospital (Unknown); Seti Zonal Hospital (Unknown); Tikapur Hospital (Unknown); Mahakali Zonal Hospital (Unknown); Bharatpur Eye Hospital (Other); B.P. Koirala Institute of Health Sciences (Other); Expertise France (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Keshab Deuba, Strategic Information Specialist, National Centre for AIDs and STD Control, Nepal
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 525; NPL-H-SCF (Other: The Global Fund to Fight AIDS, Tuberculosis and Malaria)
Record Dates: First submitted 2018-10-11; First posted 2018-10-29 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: HIV
Keywords: Package of care; Rapid Initiation of antiretroviral therapy; Advanced HIV disease; mHealth; Acquired Immunodeficiency Syndrome; Management of advance HIV disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Package of HIV care (Experimental): Screening and management (Preventive / Pre-emptive therapies dosages) of different opportunistic infections (OI), Rapid antiretroviral therapy (ART) initiation and Enhanced adherence support.
  Interventions: Combination Product: Package of HIV care
- Standard HIV care (Experimental): Screening and management of common OIs, basic health assessment (CD4, viral load and other tests), ARV drugs and follow up.
  Interventions: Combination Product: Standard HIV care

INTERVENTIONS:
Combination Product: Package of HIV care — A. Screening and management (Preventive / Pre-emptive therapies dosages) of different opportunistic infections (OI). Detail information mentioned in the manual (refer to uploaded protocol).
  B. Rapid ART Initiation
  1. PLHIV without suspicion or active OI: Initiate ART within seven days or same day after HIV serology disclosure
  2. PLHIV with suspicion or active OI: Defer initiation if clinical symptoms suggest tuberculosis or cryptococcal meningitis. Detail information mentioned in the manual (refer to uploaded protocol).
  C. Enhanced Adherence/Retention Support: mHealth: Receive text messages in mobile regarding appointment reminder (pill pick up, CD4 test, viral load test, early infant diagnosis (EID) test etc.) and general awareness messages (positive prevention, the importance of regular health check-up etc.). PLHIV with advanced HIV disease will also receive weekly/biweekly home-based adherence/ retention support linked to community care centre and community home-based care.
  Other Names: Screening and management of opportunistic infection, Rapid ART initiation and Enhanced adherence support
  Arms: Package of HIV care
Combination Product: Standard HIV care — Standard of HIV care includes screening and management of OI (OI- tuberculosis (TB), bacterial pneumonia, herpes, and candidiasis), baseline assessment (CD4 and other blood tests- complete blood count, hemoglobin, platelets, liver function test, renal function test, urine for albumin, chest x-ray), at 6 months CD4 test, viral load (twice a year) and then on a yearly basis, additional lab test at 3 months, 6 months, antiretroviral (ARV) toxicity monitoring like hemoglobin (Zidovudine), Serum Glutamic-Pyruvic Transaminase (Nevirapine/Efavirenz), Creatinine (Tenofovir), prophylaxis (Co-trimoxazole preventive therapy CD4<350 and WHO stage III and IV and Isoniazid preventive therapy if eligible) and ART / follow up (generally monthly/ bimonthly).
  Arms: Standard HIV care

SUMMARY:
This is a cluster randomized trial to determine whether a package of care including rapid antiretroviral therapy (ART) initiation, as compared to standard ART initiation, improves mortality, retention in care and viral suppression among treatment naive people living with HIV (PLHIV) in Nepal. Package of care includes immediate screening and treatment of opportunistic infections (OIs), rapid ART initiation and enhanced retention in care using mobile health (mHealth) and weekly/biweekly home-based adherence/ retention support linked to community care centre. Standard of care includes screening and management of common OIs, baseline assessment (CD4, viral load and other tests), antiretroviral drugs and ART follow up.

DETAILED DESCRIPTION:
PRAN is an open-label trial of 1000 Treatment-Naive PLHIV aged 16 years or more.

1. To evaluate whether a package of care including rapid ART initiation [diagnosis and management of opportunistic infection (OI), rapid ART initiation and enhanced adherence support] is more effective in reducing morbidity and mortality, as compared to standard ART initiation, among ART naïve PLHIV in Nepal.
2. To evaluate whether a package of care including rapid ART initiation is more effective in improving retention in HIV treatment, as compared to standard ART initiation, among ART naïve PLHIV in Nepal.
3. To evaluate whether a package of care including rapid ART initiation improves viral suppression among ART naïve PLHIV in Nepal to a higher extent than standard ART initiation,
4. To evaluate whether the different components of care act synergistically to improve mortality, retention in care and viral suppression among treatment Naive PLHIV, as compared to standard ART initiation,
5. To assess the cost-effectiveness of this package of care intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 16 years
* Diagnosed with HIV-infection
* ART-naive
* Consent for study participation

Exclusion Criteria:

* Age less than or equal to 15 years
* Any previous use of ART

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1073 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Mortality | Week 24
  All-cause mortality over the first 24 weeks after starting ART

SECONDARY OUTCOMES:
Retention in treatment | Week 48
  PLHIV alive and on ART over the first 48 weeks after starting ART
Adherence to ART | Week 0-48
  Adherence will be assessed on a monthly basis (total pills taken by patient in last month/ total pills prescribed to patient in last month).
Morbidity | Week 48
  Incidence of opportunistic infection and immune reconstitution inflammatory syndrome (IRIS)
Viral load suppression | Week 48
  PLHIV and on ART who have a suppressed viral load (<1000 copies/mL)
Cost effectiveness of Package of care | Week 48
  Intervention cost will be calculated from estimates of the per-patient quantity of services used in delivery of package of care. Cost per death prevented and cost per DALY gained.
Mortality | Week 48
  All-cause mortality over the first 96 weeks after starting ART
Hospitalization | 0-48
  Hospital inpatient episodes and total days admitted

OTHER OUTCOMES:
Cryptococcal antigen | Week 48
  Burden of serum cryptococcal antigen positive in PLHIV with CD4 < 100/mL
Immune Reconstitution Inflammatory Syndrome (IRIS) | Week 48
  Burden of IRIS
CD4 cell count | Week 48
  Changes in CD4 cell count

CONTACTS AND LOCATIONS:
Overall Officials: Basu Dev Pandey, MD, PhD, Principal Investigator — National Centre for AIDS and STD Control; Bir B Rawal, MA, Principal Investigator — National Centre for AIDS and STD Control; Rajan K Bhattarai, MPH, Principal Investigator — Save the Children; Rajya Shree Nyachhyon Kunwar, MBBS, MPH, Principal Investigator — National Centre for AIDS and STD Control/ Global Fund Programs; Upendra Shrestha, MPH, Principal Investigator — National Centre for AIDS and STD Control/ Global Fund Programs; Rajesh Khanal, MSc, Principal Investigator — National Centre for AIDS and STD Control/ Global Fund Programs; Marie Lagrange-Xelot, MD, Principal Investigator — Expertise France; Tristan Delory, MD, Principal Investigator — Expertise France; Anna Mia Ekstrom, MD, MPH, PhD, Principal Investigator — Dept of Infectious Diseases Karolinska University Hospital & Dept of Public Health (Global Health/IHCAR), Karolinska Institutet, Stockholm; Tara Nath Pokharel, MD, MPH, Principal Investigator — National Centre for AIDS and STD Control; Keshab Deuba, MMSc, PhD, Principal Investigator — National Centre for AIDS and STD Control/ Global Fund Programs
Locations (10):
- Nepal (10):
  - Sukraraj Tropical & Infectious Disease Control Hospital, Kathmandu, Bagmati
  - Bharatpur District Hospital, Bharatpur
  - Rapti Sub Regional Hospital, Dāng
  - Seti Zonal Hospital, Kailāli̇̄
  - Tikapur Hospital, Kailāli̇̄
  - Mahakali Zonal Hospital, Kañchanpur
  - National Academy of Medical Science (NAMS), Bir Hospital, Kathmandu
  - Tribhuvan University Teaching Hospital, Kathmandu
  - Western Regional Hospital, Pokhara
  - B.P. Koirala Institute of Health Sciences, Sunsari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guidelines for Managing Advanced HIV Disease and Rapid Initiation of Antiretroviral Therapy. Geneva: World Health Organization; 2017. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK475977/ PMID 29341560
- [Background] INSIGHT START Study Group; Lundgren JD, Babiker AG, Gordin F, Emery S, Grund B, Sharma S, Avihingsanon A, Cooper DA, Fatkenheuer G, Llibre JM, Molina JM, Munderi P, Schechter M, Wood R, Klingman KL, Collins S, Lane HC, Phillips AN, Neaton JD. Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection. N Engl J Med. 2015 Aug 27;373(9):795-807. doi: 10.1056/NEJMoa1506816. Epub 2015 Jul 20. PMID 26192873
- [Background] Molina JM, Grund B, Gordin F, Williams I, Schechter M, Losso M, Law M, Ekong E, Mwelase N, Skoutelis A, Wiselka MJ, Vandekerckhove L, Benfield T, Munroe D, Lundgren JD, Neaton JD; INSIGHT START study group. Which HIV-infected adults with high CD4 T-cell counts benefit most from immediate initiation of antiretroviral therapy? A post-hoc subgroup analysis of the START trial. Lancet HIV. 2018 Apr;5(4):e172-e180. doi: 10.1016/S2352-3018(18)30003-1. Epub 2018 Jan 16. PMID 29352723

DOCUMENTS (1):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03723525/Prot_000.pdf